CLINICAL TRIAL: NCT02523066
Title: Clinical Study to Evaluate the Performance of Magna Ease Heart Valve in Chinese Patients
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Magna Ease CN001
Record Dates: First submitted 2015-08-06; First posted 2015-08-14 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Mitral Valve or Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mitral Valve or Aortic Valve Replancement: One-arm group
  Interventions: Device: Magna Ease

INTERVENTIONS:
Device: Magna Ease — This study is non-intervention

SUMMARY:
Clinical Study to Evaluate the Performance of Magna Ease Heart Valve in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients who implanted with Magna Ease Heart Valve (Type:7300TFX and 3300TFX) in Fuwai Hospital in China.
* The patients agree to sign the inform consent form (ICF).

Exclusion Criteria:

* No specific exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who had the heart valves (Type: 7300TFX and 3300TFX), and are willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Echocardiography to evaluate the performance of heart valve | Up to five years after surgery
  Subjects are required to do eight times echocardiography in follow up visits

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese academy of medical sciences fuwai hospital cardiovascular disease, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.